CLINICAL TRIAL: NCT01034579
Title: A Multinational, Multicenter, Single Blood Sampling Exploratory Pharmacogenetic Study of the REGARD (the REbif® vs Glatiramer Acetate in Relapsing MS Disease) Trial
Brief Title: The REbif® vs Glatiramer Acetate in Relapsing Multiple Sclerosis Pharmacogenetics Trial
Acronym: REGARD-PGx
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: EMR200136_023
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-01

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Biomarkers; Genetic markers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rebif® Cohort (Other)
  Interventions: Other: Blood sampling
- Copaxone® Cohort (Other)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Subjects who had received Rebif® 44 microgram (mcg) three times a week for 96 weeks in study 24735 (NCT00078338) and not participated in the initial PGx sub-study will be enrolled in this retrospective cohort study wherein single blood sampling will be performed for pharmacogenetic markers analysis.
  Arms: Rebif® Cohort
Other: Blood sampling — Subjects who had received Copaxone® (Glatiramer Acetate) 20 milligram once daily for 96 weeks in study 24735 (NCT00078338) and not participated in the initial PGx sub-study will be enrolled in this retrospective cohort study wherein single blood sampling will be performed for pharmacogenetic markers analysis.
  Arms: Copaxone® Cohort

SUMMARY:
This study, REbif® vs Glatiramer acetate in relapsing multiple sclerosis (MS) disease - pharmacogenetic(s) (REGARD-PGx) is a single blood sampling exploratory pharmacogenetic study of the REGARD trial.

The aim of this trial is to provide additional data on the factors influencing interferon (IFN) beta response.

This is a Phase 4 trial involving subjects who previously participated in the REGARD trial. To address the trial objectives, a single visit follow-up trial will be performed during which a blood sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Was randomized in the REGARD 24735 study
* Is willing and able to comply with the protocol
* Has given written informed consent before performing any trial-related activities

Exclusion Criteria:

* Is unwilling or unable to participate in the study
* Is already included in the initial REGARD 24735 PGx sub-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Verdun di Cantogno, MD, Study Director — Merck Serono S.A., Geneva
Locations (1):
- Please Contact U.S. Medical Information Located in, Rockland, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 758 participants randomized and treated in study 24735 (NCT00078338), 326 were enrolled in EMR200136_023 (NCT01034579) out of which 2 participants, who had participated in initial pharmacogenetics (PGx) sub-study, were found to be ineligible and therefore, evaluable population for EMR200136_023 (NCT01034579) comprised of 324 participants.
Groups:
- Rebif® Cohort: Participants who had received Rebif® 44 microgram (mcg) three times a week for 96 weeks in study 24735 (NCT00078338) and not participated in the initial PGx sub-study were enrolled in this retrospective cohort study wherein single blood sampling was performed for pharmacogenetic markers analysis.
- Copaxone® Cohort: Participants who had received Copaxone® (Glatiramer Acetate) 20 milligram once daily for 96 weeks in study 24735 (NCT00078338) and not participated in the initial PGx sub-study were enrolled in this retrospective cohort study wherein single blood sampling was performed for pharmacogenetic markers analysis.
Period: Overall Study
Arm/Group | Rebif® Cohort | Copaxone® Cohort
Started | 158 | 166
Completed | 158 | 166
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Evaluable population included all randomized participants who had received at least 1 dose of Rebif® or Copaxone® in 24735 (NCT00078338) and not participated in the initial PGx sub-study and provided consent to take part in this EMR200136_023 study (NCT01034579).
Groups:
- Rebif® Cohort: Participants who had received Rebif® 44 microgram (mcg) three times a week for 96 weeks in study 24735 (NCT00078338) and not participated in the initial pharmacogenetics (PGx) sub-study were enrolled in this retrospective cohort study wherein single blood sampling was performed for pharmacogenetic markers analysis.
- Total: Total of all reporting groups
Arm/Group | Rebif® Cohort | Copaxone® Cohort | Total
Number analyzed (Participants) | 158 | 166 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (9.5) | 37.4 (9.5) | 36.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 119 | 218
  Male | 59 | 47 | 106

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders as Defined by Single Nucleotide Polymorphism (SNP) Markers
Description: A responder was defined as a participant with no multiple sclerosis (MS) relapse and no Expanded Disability Status Scale (EDSS) progression during 96 weeks in 24735 (NCT00078338). All responders were categorized on the basis of following six SNP markers: SNP1, SNP2, SNP3, SNP4, SNP5, and SNP6. Two types of variables were possible for each SNP marker: two-level genotype-based or three-level allele-based association variables. For the two-level genotype-based SNP markers (SNP2, SNP4, and SNP6), the absence or presence of the genotype was analyzed as the dichotomous variable as 0 (absence of the genotype) and 1 (presence of the genotype). For the three-level allele-based association SNP markers (SNP1, SNP3, and SNP5), the analysis was based on the number of copies of the allele (0, 1 and 2). Percentage of responders segregated on the basis of SNP marker variable were reported.
Time Frame: Day 1 of EMR200136_023 study
Population: Evaluable population. Here, 'N' signifies number of participants who were evaluable for this outcome measure and 'n' signifies number of participants who were evaluable for the specified SNP categories.
Measure: Number; unit: percentage of participants
Arm/Group | Rebif® Cohort | Copaxone® Cohort
Number analyzed (Participants) | 135 | 149
percentage of participants
  SNP1: 0 copy (n=63, 61) | 63.5 | 63.9
  SNP1: 1 copy (n=61, 73) | 65.6 | 60.3
  SNP1: 2 copies (n=11, 15) | 72.7 | 73.3
  SNP2: Present (n=106, 121) | 61.3 | 64.5
  SNP2: Absent (n=29, 28) | 79.3 | 57.1
  SNP3: 0 copy (n=62, 72) | 67.7 | 65.3
  SNP3: 1 copy (n=64, 62) | 60.9 | 56.5
  SNP3: 2 copies (n=9, 15) | 77.8 | 80.0
  SNP4: Present (n=73, 77) | 63.0 | 61.0
  SNP4: Absent (n=62, 72) | 67.7 | 65.3
  SNP5: 0 copy (n=58, 66) | 65.5 | 60.6
  SNP5: 1 copy (n=54, 67) | 64.8 | 67.2
  SNP5: 2 copies (n=23, 16) | 65.2 | 56.3
  SNP6: Present (n=18, 27) | 55.6 | 63.0
  SNP6: Absent (n=117, 122) | 66.7 | 63.1

2. Secondary Outcome: Number of Participants With Confirmed Expanded Disability Status Scale (EDSS) Progression as Defined by SNP2 Marker
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. EDSS progression was defined as increase by at least 1 point if last value of EDSS was equal to 5.5, and by at least 0.5 points if last EDSS was more than 5.5. SNP2 is two-level genotype-based SNP marker. The absence or presence of the genotype was analyzed as the dichotomous variable as 0 (absence of the genotype) and 1 (presence of the genotype). Number of responders segregated on the basis of SNP2 marker variable were reported.
Time Frame: Day 1 of EMR200136_023 study
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Rebif® Cohort | Copaxone® Cohort
Number analyzed (Participants) | 135 | 151
participants
  SNP2: Present (n=106, 123) | 16 | 16
  SNP2: Absent (n=29, 28) | 3 | 0

3. Secondary Outcome: Change in Time Constant 1 Gadolinium (T1 Gd) Enhancing Lesion Volume as Defined by SNP3 and SNP4 Markers
Description: Change in T1 Gd enhancing lesion volume was measured by using magnetic resonance imaging (MRI) scans. SNP4 is two-level genotype-based SNP marker. The absence or presence of the genotype was analyzed as the dichotomous variable as 0 (absence of the genotype) and 1 (presence of the genotype). SNP3 is a three-level allele-based association SNP markers. The analysis was based on the number of copies of the allele (0, 1 and 2). Change in T1 Gd enhancing lesion volume segregated on the basis of SNP3 and SNP4 marker variables were reported.
Time Frame: Baseline (Day 1 of 24735 [NCT00078338] study) and Day 1 of EMR200136_023 study
Population: MRI evaluable population was defined to include all participants from the evaluable population who had at least one post-baseline MRI evaluation during study 24735. Here, 'N' signifies number of participants who were evaluable for this outcome measure and 'n' signifies number of participants who were evaluable for the specified SNP categories.
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Rebif® Cohort | Copaxone® Cohort
Number analyzed (Participants) | 65 | 69
cubic millimeter (mm^3)
  SNP3: 0 copy (n=30, 42) | -524.23 (1481.03) | -203.71 (687.59)
  SNP3: 1 copy (n=31, 22) | -106.97 (152.22) | -61.95 (232.25)
  SNP3: 2 copies (n=4, 5) | -26.50 (53.00) | -22.80 (34.27)
  SNP4: Present (n=35, 27) | -97.77 (146.18) | -54.70 (209.73)
  SNP4: Absent (n=30, 42) | -524.23 (1481.03) | -203.71 (687.59)

4. Secondary Outcome: Change in Brain Volume as Defined by SNP2 Marker
Description: Change in brain volume was measured as the brain parenchymal fraction using MRI scans. SNP2 is two-level genotype-based SNP marker. The absence or presence of the genotype was analyzed as the dichotomous variable as 0 (absence of the genotype) and 1 (presence of the genotype). Change in brain volume segregated on the basis of SNP2 marker variables were reported.
Time Frame: Baseline (Day 1 of 24735 [NCT00078338] study) and Day 1 of EMR200136_023 study
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Rebif® Cohort | Copaxone® Cohort
Number analyzed (Participants) | 44 | 44
cubic millimeter (mm^3)
  SNP2: Present (n=33, 38) | -1.51 (1.60) | -1.10 (1.16)
  SNP2: Absent (n=11, 6) | -0.57 (1.25) | -0.48 (0.41)

5. Secondary Outcome: Mean Number of Time Constant 2 (T2) Active Lesions Per Subject Per Scan as Defined by SNP5 Marker
Description: Mean number of T2 active lesions was measured by using MRI scans. SNP5 is a three-level allele-based association SNP markers. The analysis was based on the number of copies of the allele (0, 1 and 2). Mean number of T2 active lesions segregated on the basis of SNP5 marker variables were reported.
Time Frame: Day 1 of EMR200136_023 study
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T2 lesions
Arm/Group | Rebif® Cohort | Copaxone® Cohort
Number analyzed (Participants) | 78 | 83
T2 lesions
  SNP5: 0 copy (n=31, 42) | 0.72 (1.50) | 1.05 (1.32)
  SNP5: 1 copy (n=36, 34) | 0.53 (1.41) | 0.55 (1.19)
  SNP5: 2 copies (n=11, 7) | 0.30 (0.40) | 0.18 (0.37)

ADVERSE EVENTS:
Description: As it is a retrospective study, only serious adverse events which were considered by the investigator to be at least possibly related to the conduct of the trial, that is, the trial procedure (blood sampling), were collected.
Arm/Group | Rebif® Cohort | Copaxone® Cohort
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/166
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs have to submit any publication for internal review and approval by EMD Serono before it can be publicly disclosed.